CLINICAL TRIAL: NCT04845607
Title: Prophylactic Amiodarone for Shockable Cardiac Arrest During Targeted Post Cardiac Arrest Care: Multi-center, Open Labelled Randomized Controlled Trial
Brief Title: Prophylactic Amiodarone for Shockable Cardiac Arrest
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Won Young Kim (Other)
Responsible Party: Sponsor-Investigator, Won Young Kim, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PASCA trial
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Arrest; Ventricular Arrythmia
MeSH Terms: conditions — Heart Arrest | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic amiodarone (Experimental)
  Interventions: Drug: Amiodarone Injection
- Conventional management (No Intervention)

INTERVENTIONS:
Drug: Amiodarone Injection — Amiodarone continuous infusion during 24 hours from return of spontaneous circulation.
  Arms: Prophylactic amiodarone

SUMMARY:
The aim of this study is to determine whether the prophylactic amiodarone can prevent re-arrest with ventricular shockable rhythm in patients who treated with targeted temperature management after return of spontaneous circulation from cardiac arrest which had been shockable rhythm during CPR.

DETAILED DESCRIPTION:
Patients with cardiac arrest are in high risk of re-arrest during post cardiac arrest care due to vulnerable heart state electrically and hemodynamically. Especially if patients who had experienced shockable rhythms such as ventricular fibrillation or pulseless ventricular tachycardia during CPR, then they are at high risk of developing shockable re-arrest.

However until now there has not been any evidence of prophylactic anti arrhythmic drug effect during post cardiac arrest care.

Amiodarone is class III anti arrhythmic drug which has been used for conversion of ventricular arrhythmia during CPR.

In this study we want to determine whether the prophylactic amiodarone can prevent re-arrest with ventricular shockable rhythm or not.

ELIGIBILITY:
Inclusion Criteria:

* Non traumatic cardiac arrest patients who had VF or pVT during CPR in ER

Exclusion Criteria:

* age < 18 yr
* pregnancy
* non cardiac caused arrest such as hanging
* previous amiodarone continuous infusion before radomization
* sustained ventricular arrhythmia recurrence after ROSC
* extracorporeal membrane oxygenation
* contra indication for amiodarone
* disagree with this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients with re-arrest by shockable rhythm | 5 days from return of spontaneous circulation
  No recurrence of ventricular fibrillation or pulseless ventricular tachycardia

OTHER OUTCOMES:
3 month survivor | 3 months after the time of hospital discharge
  mortality
3 months neurological outcome | 3 months after the time of hospital discharge
  cerebral performance scales 3, 4 and 5

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No